CLINICAL TRIAL: NCT03720873
Title: An Multicenter,Phase II Trial of EGFR-TKIs Combine With Anlotinib as First-line Treatment for Patients With Advanced EGFR Mutation-positive NSCLC
Brief Title: EGFR-TKIs Combine With Anlotinib as First-line Treatment for Patients With Advanced EGFR Mutation-positive NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: secgolc004
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: EGFR Gene Mutation
MeSH Terms: interventions — Erlotinib Hydrochloride; Gefitinib; icotinib; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EGFR-TKIs and Anlotinib (Experimental): Experimental:EGFR-TKIs and Anlotinib EGFR-TKIs:erlotinib 150mg QD or gefitinib250mgQD or icotinib 125 mg TID , Anlotinib 12mg po qd d1-14 q21d
  Interventions: Drug: erlotinib or gefitinib or icotinib; Drug: Anlotinib

INTERVENTIONS:
Drug: erlotinib or gefitinib or icotinib — Patients will be treated with erlotinib 150mgQD or gefitinib250mgQD or icotinib 125 mg TID
Drug: Anlotinib — Patients will be treated with Anlotinib 12mg po d1-14 Q21d

SUMMARY:
A single arm study: EGFR-TKIs Combine With Anlotinib as First-line Treatment in patients with EGFR-mutant non-small-cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This trial investigated the efficacy and safety of EGFR-TKIs Combine With Anlotinib as First-line Treatment in patients with EGFR-mutant NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 18 years
* ECOG performance status 0-1
* Adequate haematological function, coagulation, liver function and renal function
* Pathological diagnosis of predominantly non-squamous, non-small-cell lung cancer (NSCLC)
* TNM version 7 stage IV disease including M1a (malignant effusion) or M1b (distant metastasis), or locally advanced disease not amenable to curative treatment (including patients progressing after radiochemotherapy for stage III disease)
* Measurable or evaluable disease (according to RECIST 1.1 criteria).
* Centrally confirmed EGFR exon 19 deletion (del19) or exon 21 mutation (L858R)

Exclusion Criteria:

* - Patients who have had in the past 5 years any previous or concomitant malignancy EXCEPT adequately treated basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix or bladder, in situ breast carcinoma.

Patients with any known significant ophthalmologic anomaly of the ocular surface

* Patients who received prior chemotherapy for metastatic disease
* CNS metastases
* Patients who received previous treatment for lung cancer with drugs targeting EGFR or VEGF
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | within 6 months of the last visit of last patient, approximately 30 months after inclusion of first patient
  Time from the date of enrolment to discontinuation of treatment for any reason (including progression of disease, treatment toxicity, refusal and death)

SECONDARY OUTCOMES:
Objective response | through study completion,an average of three years
  Best overall response (complete remission or partial remission) across all assessment time-points according to RECIST Criteria 1.1, during the period from enrolment to termination of trial treatment.
Safety - Adverse events graded according to NCI CTCAE V4.03 | within 6 months of the last visit of last patient, approximately 30 months after inclusion of first patient
  Adverse events graded according to NCI CTCAE V4.03
Overall survival | Three years
  Defined as the time in month from diagnosis of recurrent NPC to the date of death is observed or to last follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong He, master, Principal Investigator — Fujian Cancer Hospital
Locations (1):
- Fujian cancer hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external indepentent Review Panel. Requesdtors will be required to sign a Data Access Agreement.

REFERENCES:
- [Result] Maemondo M, Fukuhara T, Sugawara S, et al. NEJ026: Phase III study comparing bevacizumab plus erlotinib to erlotinib in patients with untreated NSCLC harboring activating EGFR mutations[J]. Annals of Oncology, 2016, 27